CLINICAL TRIAL: NCT05441137
Title: Using Head-mounted, Eye-tracking to Compare Looking, Manual Exploration and Social Interaction During Active Locomotion in Toddlers With Mild, Moderate and Severe Motor Delays: A Randomized Controlled Trial
Brief Title: Using Head-mounted, Eye-tracking to Compare Looking, Manual Exploration and Social Interaction During Active Locomotion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiang-Han Huang, Associate Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111WFD2610060
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Young Children With Motor Disabilities
MeSH Terms: interventions — Sitting Position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A ROC with a Standing Posture for Toddlers with Mild Motor Delays (ROC-Stand(Mild)) (Active Comparator): The whole study duration will be 24 weeks, including a 12-week intervention and a 12-week follow-up. All programs will include 120 minutes/per session, 2 sessions/per week. Each week the research team will help the participant wear a wireless, head-mounted eye-tracker (46g) for recording the first 20-minute of both driving and natural play sessions in a 2-hour training session. The 2-hour training session is composed of a 70-minute driving session and a 40-to-50-minute natural play session, with a 10-mintue break if necessary according to the previous ROC-related studies. The natural play session can be divided into two 20-to-25-minute sessions depending on the participant's condition. The head-mounted cameras worn by the participants and caregivers will record the visual and manual behaviors for 40 minutes/per week during intervention. All programs will be discussed by the family, the treating therapist and the research team.
  Interventions: Behavioral: Ride-On Cars Training with Different Postures
- A ROC with a 25-minute Standing Posture for Children with Moderate Motor Delays (ROC-Stand25(Mod)) (Active Comparator): The training guidelines and time are the same as the ROC-Stand(Mild) group, except for the participant's severity level of motor delay and using a 25-minute standing and 45-mnute sitting posture for driving. The participants will also wear the head-mounted eye tracker in one training session every week.
  Interventions: Behavioral: Ride-On Cars Training with Different Postures
- A ROC with a Sitting Posture for Children with Severe Motor Delays (ROC-Sit(Sev)) (Active Comparator): The training guidelines and time are the same as the ROC-Stand(Mild) group, except for the participant's severity level of motor delay and using a sitting posture for driving. The participants will wear the head-mounted eye tracker in one training session every week.
  Interventions: Behavioral: Ride-On Cars Training with Different Postures
- Conventional Therapy for Children with Mild Motor Delays (Control(Mild)) (Placebo Comparator): The whole study duration will be 24 weeks, including a 12-week intervention and a 12-week follow-up. All programs will include 120 minutes/per session, 2 sessions/per week. Each participant will have the opportunity to walk on certain public space as the ROC training groups and interact with the therapist and caregivers depending on his/her motor abilities. The participants will also wear the head-mounted eye-tracker in one training session every week.
  Interventions: Behavioral: Conventional Therapy
- Conventional Therapy for Toddlers with Moderate Motor Delays (Control(Mod)) (Placebo Comparator): The training guidelines and time are the same as the Control(Mild) group, except for the participant's severity level of motor delay. The participants will wear the head-mounted eye-tracker in one training session every week.
  Interventions: Behavioral: Conventional Therapy
- Conventional Therapy for Toddlers with Severe Motor Delays (Control(Sev)) (Placebo Comparator): The training guidelines and time are the same as the Control(Mild) group, except for the participant's severity level of motor delay. The participants and caregivers will also head-mounted eye-tracker in one training session every week.
  Interventions: Behavioral: Conventional Therapy

INTERVENTIONS:
Behavioral: Ride-On Cars Training with Different Postures — A licensed, independent therapist and caregivers will provide the training program in the public space in the university for a total of 12-week intervention based on ecological and dynamic systems theories. Training will concentrate on building the concept of casual-effect on the control system and car motion, practicing goal-oriented driving (e.g., driving 200 meters and reach for a toy or contact with a person, play hide-and-seek) in certain public spaces, including hallways, convenient stores, garden, museum and upper limb use in functional tasks with driving, facilitating hand use in functional tasks for exploration and applying various motor skills for mobility and socialization in natural play session. Every week's treatment program will preplanned and adjusted by the therapist and the caregivers through discussion and clinical observation of participant's performance in the previous session. Participants will continue their regular therapy during the whole study.
  Other Names: Ride-On Cars with Standing Postures; Ride-On Cars with 25-min Sitting and 45-min Standing Postures; Ride-On Cars with Sitting Postures
  Arms: A ROC with a 25-minute Standing Posture for Children with Moderate Motor Delays (ROC-Stand25(Mod)); A ROC with a Sitting Posture for Children with Severe Motor Delays (ROC-Sit(Sev)); A ROC with a Standing Posture for Toddlers with Mild Motor Delays (ROC-Stand(Mild))
Behavioral: Conventional Therapy — The other independent OT will be responsible for providing conventional therapy based on the developmental and motor learning theories. The goals are to improve certain motor skills or psychosocial skills based on each participant's current developmental stage. The general propose of the training is to facilitate the developmental scales and improve mobility, socialization and upper limb use in functional tasks.
  Arms: Conventional Therapy for Children with Mild Motor Delays (Control(Mild)); Conventional Therapy for Toddlers with Moderate Motor Delays (Control(Mod)); Conventional Therapy for Toddlers with Severe Motor Delays (Control(Sev))

SUMMARY:
The three purposes of this study are: 1) to determine the feasibility of using a head-mounted eye-tracker and examine the effects of the optimal mobility training on increasing visual and manual exploration in toddlers with different severity levels of motor delays, 2) to compare the effectiveness of providing optimal mobility training on outcomes across the ICF framework in toddlers with mild, moderate and severe motor delays, and 3) to determine the effects of optimal mobility training on the relationship among looking and manual actions, caregiver-child interactions and mastery motivation in toddlers with mild, moderate and severe motor delays.

Based on the power analysis from the preliminary results of the pilot study, we will recruit 72 toddlers with motor delays and further assign them to the mild, moderate or severe motor delays group. The participants in each group will be randomly assigned to either the ROC training program or conventional therapy (Control) program, resulting the following six training groups: the ROCStand(Mild) group (n=12), the ROC-Stand25(Mod) group (n=12), the ROCSit(Sev) group (n=12), Control(Mild) group (n=12), Control(Mod) group (n=12), and Control(Sev) group (n=12). The whole study duration will be 24 weeks, including a 12-week intervention and a 12-week follow-up. All programs will include 120 minutes/per session, 2 sessions/per week. Participants will continue their regular therapy during the whole study. The head-mounted cameras worn by the participants and caregivers will record the visual and manual behaviors for 40 minutes/per week during intervention. Standardized assessments are provided for a total three times, including the time before and after the intervention and in the end of the follow-up phase. Assessments include body function, mobility, psychosocial function, family perception and participation. The findings of this study will provide guidelines for arranging the training environment depending on each child's and family's needs.

DETAILED DESCRIPTION:
Although environmental and task modifications are powerful methods used to affect function in rehabilitation and frequently used by the therapists, these modifications are typically introduced using a trial and error approach. A better understanding of the fits between the child and the environment may help therapists develop a more structured approach to manipulating environmental and task characteristics in order to enhance the emergent actions of children. The important factors required to achieve positive effects of ride-on car (ROC) training include the"fit"between a child's characteristics, the modified ROC, and the physical and social contexts.

Based on the findings of previous randomized controlled trials (RCTs) (NCT03707405), children with mild motor delay may gain the most from using the ROC-Stand style for 70 minutes (ROC-Stand) while those with moderate motor delay may gain the most with a 25-minute standing posture and a 45-minute sitting posture (ROC-Stand25). Children with severe motor delay may benefit more from the ROC training in a sitting posture (ROC-Sit), which may provide moderate challenges as an optimal mobility training program. Thus, the heterogeneity of the participants regarding severity level of motor delays and environmental considerations may be the factors contributing to the different treatment effects.

A new technical challenge occurs to record and capture young children's visual and haptic exploration. Infants cannot attend to the entire visual field captured by the action camera and their attention constantly shifts between areas of the visual field. It is difficult to differentiate what the targets the child actually fixates at or interacts with. To allow the direct observation of infants' spontaneous eye movements during self-initiated locomotion, Dr. Adolph have used a wireless, head-mounted eye-tracker (Positive Science, LLC) which could measure infants' visual behaviors during free, unfettered locomotion. This novel methodology includes a lightweight and comfortable headgear, transmitter, and battery pack which can record infants' eye gaze. The analysis can focus on where infants look during self-initiated locomotion, object exploration and in response to caregivers' vocalizations. The combination of the ROC training with this head-mounted eye-tracker will allow us to further track what visual and haptic information is obtained during the early PMD use. It is helpful for understanding the influences of environmental factors on psychosocial function in toddlers with motor delays.

To provide a full investigation of the effectiveness of optimal mobility training, this study proposes to compare the effects on toddlers with mild, moderate and severe motor delays. Additionally, a wireless, head-mounted eye-tracker will be applied as the novel method to analyze children's looking, manual behaviors and social interaction during the training phase.

The specific aims of this study are: 1) to determine the feasibility of using a head-mounted eye-tracker and examine the effects of the optimal mobility training on increasing visual and manual exploration in toddlers with different severity level of motor delays, 2) to compare the effectiveness of providing optimal mobility training on outcomes across the ICF framework in toddlers with mild, moderate and severe motor delays, and 3) to determine the effects of optimal mobility training on the relationship among looking and manual actions, caregiver-child interactions and mastery motivation in toddlers with mild, moderate and severe motor delays.

Method Study Design: A multiple pretest-posttest control group design will be applied. On the basis of our previous pilot findings in toddlers with mild, moderate and severe motor delays, 6 groups will be involved in this project: using a ride-on car in a standing posture for driving for children with mild motor delay (ROC-Stand(Mild)), conventional therapy for those with mild delay (Control(Mild)), a 25-minute standing posture and 45-minute sitting posture for driving for those with moderate motor delay (ROC-Stand25(Mod)), conventional therapy for those with moderate delay (Control(Mod)), a sitting posture for those with severe motor delay (ROC-Sit(Sev)), and conventional therapy for those with severe delay (Control(Sev)). Based on the previous RCTs, the study duration for each participant is 24 weeks, including a 12-week training phase (intervention) and a 12-week follow-up phase.

Participants: 72 participants aged 12 months to 36 months old with motor delays will be recruited in the study and determined the severity level of motor delays based on the cutoff values of Bayley-III MC scores (mild: 70-84; moderate: 55-69; severe: <55). 24 toddlers with mild motor delays will be in one group, 24 toddlers with moderate motor delays in another group and the other group has 24 toddlers with severe motor delays. Participants in each group will be randomly assigned to a ROC training group or conventional therapy (Control) group. There will be 6 groups, including the ROC-Stand(Mild) group (12 toddlers), the Control(Mild) group (12 toddlers), the ROC-Stand25(Mod) group (12 toddlers), the Control(Mod) group (12 toddlers), ROC-Sit(Sev) group (12 toddlers) and Control(Sev) group (12 toddlers).

Recruitment: The participants will be recruited from self-referrals, health care practitioners, or the hospitals in Taipei or Taoyuan where toddlers with motor delays are receiving outpatient rehabilitations. The research team will initially post flyers describing the study at clinical settings and contact the therapists in the clinical settings to introduce the goals, criteria and general procedure of the study. Parents/guardians will obtain information about the study through the flyers and their therapists. The research team will contact the parent/guardian to explain study details and provide them the opportunity to ask questions. Children of parents/guardians who provide informed consent will participate in the study.

Procedure: Before randomization, the participants will receive pre-intervention measurements, including standardized assessments of developmental abilities, the evaluations of environmental factors and parental-perception questionnaires. An independent, licensed OT or PT who is blinded to the study purpose and not involved in the training programs will complete the pretest and posttest assessments and questionnaires in a testing room at Chang Gung University. These assessments will occur on three occasions: before and after the 12-week training phase, i.e., intervention (T1 & T2) and the end of the 12-week follow-up phase (T3). After the pretest, participants are arranged to the group of mild motor delays, moderate motor delays or severe motor delays based on the cutoff values of Bayley-III MC scores. After allocation, participants will be randomly assigned into the ROC training or conventional therapy groups, resulting in 6 groups. All the participants will start the training programs in a training room and certain public space in the university. During the 12-week intervention, the locomotor experience of eye gaze and the accompanying manual actions, and social interactions for the 6 training groups will be recorded by a wireless, head-mounted eye-tracker worn by the participants for one 2-hour session/per week at the university. An activity log used in the previous studies will also be applied to record the training conditions and the caregiver's feedback on the training programs every week during the 12-week intervention. The activity log will be mostly qualitative data that involves caregivers' descriptions. For the 12-week follow-up phase, all participants will not receive any training program from the research team. They only have their regular therapy from their own hospitals or clinics. The information of regular therapy, including the type, the frequency and the dosage, will be collected at T1, T2 and T3.

Intervention: The therapists who only involve providing the training programs will ask caregivers to identify goals and measure progress using goal attainment scaling (GAS) at T1, T2 and T3 time points for the 6 groups. Two independent licensed therapists (OT or PT) who will not involve the administration of assessments will provide the ROC training or conventional therapy programs, respectively. One training provider is responsible for the ROC-related programs which require the therapist working with the caregivers based on the coaching technique described in the FCS model. The ROC involves a standing, a combined or a sitting posture depending on their severity level of motor delays. The training principles are similar to those applied in the previous studies of ROC training in various environments. The other therapist is responsible for the conventional therapy which is a child-centered, therapist-directed program. Participants will have a necessary break depending on their endurance during training. In addition, all participants in the 6 groups will wear the eye-tracking headgear to record the looking, manual and interactive behaviors for one session/per week during intervention. All participants in the 6 groups will continue their regular therapy from their own hospitals or clinics throughout the 24-week duration of the study, including physical therapy, occupational therapy, and speech therapy.

Follow-up: This period will involve a 12-week phase following the above treatment programs; during this time no treatment programs will be delivered to the participants except for their own regular therapy.

Instrument and Procedure: To obtain the data of locomotor experience, an objective measure of a head-mounted, eye-tracker and a qualitative measure of activity logs will be applied during the 12-week intervention phase. Standardized assessments as the quantitative measures across the ICF framework will be administered at T1, T2, and T3 in a testing room of the university.

Descriptive statistics (frequency, means, standard deviations) of each behavior will be calculated. Kolmogorov-Smirnov will be used to examine whether the data follows a normal distribution. To compare the baseline characteristics of the major 3 groups categorized as mild, moderate and severe motor delays, one way ANOVA (for data with normal distribution) and Kruskal-Wallis analysis of variance (for data with non-normal distribution) will be conducted. Data will be analyzed based on an intention-to-treat analysis. For those data collected during the 12-week intervention, descriptive statistics (frequency, means, standard deviations) of looking, manual actions and interactive behaviors will be calculated and repeated measures analysis of variance (group [6] × time [12]) will be used to compare the effects on each exploratory behaviors among the 6 training groups during intervention. A repeated measures analysis of variance (group [6] × time [3]) will be employed to evaluate the treatment effects on the secondary outcomes within and among the 6 groups at T1, T2, and T3, followed by a post-hoc analysis using Bonferroni test to determine between which groups the differences occur. To clarify the relationship between other relevant factors and psychosocial outcomes, we will consider two co-variates in the analysis based on previous research: MC scores from the Bayley-III and caregiver-child dysfunctional interaction (obtained from PSI). Last, we will apply a coefficient test for analyzing the relationship among the social function, looking/manual actions and social interactions, and mastery motivation during the intervention phase in each group. The scores of social function and mastery motivation will be based on the mean change scores from T1 to T2. The mean frequency of total looking/manual actions and social interactions will be calculated from the coding results of the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

1. motor delays that resulted in motor impairments preventing independent walking (standard deviation [SD] <-1.5, assessed by the Chinese Child Development Inventory via a pediatric physician)
2. being able to stand independently for two seconds or tolerate standing with support for 10 minutes
3. being able to reach objects with either one or both hands
4. 69 to 103 cm height and 7 to 18 kg weight
5. parents agreeing to provide consent for their child's participation in the training program

Exclusion Criteria:

1. children with severe sensory impairments (including blindness or deafness)
2. exceeding the height or weight criteria
3. parents/guardians who were unable to make the time commitment for the program and children with severe emotional disorders resulting in strong reactions and causing possible harms.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Face Looking | 40-minute each week during the intervention phase
  The frequency (number of times) and duration (in seconds) that the child looks at the interacting person (social partner). Looking at the face will be scored any time if the circular cursor contains any part of the social partner's face, between the chin and the hairline; hair and the back of the head are not included. Additionally, we assume participants' gaze to be directed at the social partner's face if both the gaze location and the face are above the boundary of the video frame.
Body Looking, Toy and Environment Looking | 40-minute each week during the intervention phase
  The frequency (number of times) and duration (in seconds) that the child looks at the person's body or toy. Looking at bodies will be scored when the circular cursor intersects with any part of the body, excluding the face. In addition, body looking is also scored if the gaze cursor falls on a toy held in the hands of the social partner. Body looking includes all person-directed looking except face looking. Looking at the toys is scored any time when the circular cursor contains any part of the toys and does not contain the partner's face. The same video can be counted as both toy and body looking if looking is directed at a toy held by the caregiver. Environment looking includes all looking except face, body and toy looking. Looking at the environment is scored any time when the circular cursor contains any part of an object or physical structure of the environment, e.g., wall, door, floor, box…etc.
Visual Fixations during Obstacle Encounter | 40-minute each week during the intervention phase
  The frequency (number of times) and duration (in seconds) of fixations will be coded. Obstacle encounter refers to the child's PMD or leading limb contacts the new surfaces, e.g., up, down or over a surface of a different height or texture. Coders will identify fixations in the 5 seconds prior to obstacle encounter. An obstacle fixation is counted if the gaze crosshair rests stably on the obstacle for 3 or more consecutive frames (100ms). We will score any fixation within a car's or step's length of where children actually drive or place their limbs. If the child fixates the surface multiple times in the 5 seconds period, we will only count the fixation occurs closest moment of the encounter. Fixation initiation will be scored from the start of the fixation until the moment of the encounter. Fixation termination will be scored from the last frame of that fixation until the moment of the encounter.
Visual Fixations during Manual Encounter | 40-minute each week during the intervention phase
  The frequency (number of times) and duration (in seconds) will be coded. Manual encounter refers to the child's hand contacts the objects or toys. We will only count the first object touch during repetitive bouts during which touches of the same object occur within 2 seconds of each other. For each manual encounter, we will score object fixations in the 5 seconds prior to contacting the object with the hand. Because objects may be in motion before the child reaches for them, we will include both fixations and smooth pursuit of objects, provided gaze is stable on the target for 100 ms. We will only count the last fixation before the manual encounter in the event of multiple fixations or smooth pursuits.
Social Encounter | 40-minute each week during the intervention phase
  The frequency (number of times) and duration (in seconds) will be coded. Social encounter refers to the social partner's any speech sound directs toward the child separated by at least 0.5 seconds from the previous vocalization. We will code each time that the child fixates his/her social partner, including face, hands, or body.
Fixations to Destinations | 40-minute each week during the intervention phase
  The frequency (number of times) and duration will be coded. Fixations will be counted if the destination is within the 4°gaze indicator for three consecutive frames (~90 ms). Locomotion ending at destinations are destination directed if the child fixates the destination during the period between the last destination and the current locomotion initiation. Discovery locomotion occurs when the child travels to a new destination that is fixated after the child is already in motion, or if the child stops moving near a destination that is never fixated.

SECONDARY OUTCOMES:
The Bayley Scales of Infant and Toddler Development-Third Edition (Bayley-III) | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  An internationally recognized set of developmental tests with high reliability and validity applied to examine participants' developmental abilities. The Bayley has subsets of tests for motor, cognitive, and language development for children aged from 1 month to 42 months. It is a standardized assessment that can classify children's severity level of motor delays into four levels based on their motor composite scores, classified as severe (scores <55), moderate (55-69), mild (70-84), and no (>85) motor delays.
Infant/Toddler Sensory Profile - Chinese version (ITSP-C) | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  A standardized, norm-reference questionnaire of sensory processing ability in children at 0-3 years of age from caregiver's observations. Based on the criteria of age, the version for older children (7-36 months old) consisting of 48 item questions will be used in this study. The ITSP-C includes five sensory processing sections (Auditory, Visual, Vestibular, Tactile, and Oral Sensory Processing) and uses a 5-point Likert scale from 1 (almost always) to 5 (almost never). The ITSP-C with the Taiwanese norm has been established with good reliability and validity.
Peabody Developmental Motor Scales - Second edition (PDMS-2) | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  A norm referenced, standardized assessment of gross and fine motor skills in children 0-6 years. The PDMS-2 has been validated as a discriminative measure and demonstrated its' responsivity to change in infants and toddlers with cerebral palsy.
The Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  A caregiver's report questionnaire and five-point scale which measures both the instrumental and expressive aspects of mastery motivation. The DMQ involves seven subscales, including cognitive/object persistence, gross motor persistence, social mastery motivation with adults, social mastery motivation with children/peers, mastery pleasure, negative reactions to challenge in mastery situations, and general competence. A higher score indicates higher motivation. For children aged 6 months to 19 years, the DMQ 18 previously showed good validity and reliability. Considering the age of participants, this study used two versions of the DMQ 18: infant's version (6-18 months) and preschooler's version (1.5-5 years).
The Chinese version of Pediatric Evaluation of Disability Inventory (PEDI-C) | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  A set of tests for children from 8 months to 6 years old. The PEDI-C quantifies self-care, mobility, and social function, and is particularly useful for tracking changes in functional skills. Each domain can be used separately for data analysis. The inter-rater and intra-rater reliabilities of the study reveal excellent agreement of the observations (0.95-0.99), and good concurrent validity with the Functional Independence Measure for Children (Spearman ρ, 0.92-0.99).
Goal Attainment Scale (GAS) | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  A family-centered, criteria-referenced, responsive tool that includes five possible outcomes. A score of 0 indicates that the child has attained the goal, scores of -2 and -1 represent lower than expected performance, and +1 and +2 are higher than expected performance. It had good validity and excellent inter-rater agreements with ICCs of 0.90 or higher. The goals were incorporated into a single GAS composite score and converted to a T-score. A mean T-score of 50 indicated that the participants exceeded the expected level of goal performance.
The Chinese version of the Affordance in the Home Environment for Motor Development - Toddler version (AHEMD-Toddler-C) | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  A reliable and valid assessment to assess the quality and quantity of motor development opportunities in the home during early childhood. Age-related AHEMD questionnaires were developed (3-to-18 months; and 18-to-42 months) and translated into four different languages: English, Chinese, Portuguese, and Spanish. Test-retest reliabilities for AHEMD-Toddler-C were adequate (0.46~0.93); for convergent validity, the correlation coefficients between AHEMD and HOME were 0.44.
The Parenting Stress Index Short Form (PSI/SF) | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  A tool to measure measures the overall level of parenting stress experienced by parents/caregivers of children aged between one month and 12 years. The three subscales, that is, parental distress, parent-child dysfunctional interaction, and difficult child, add up to a total stress score. A higher score indicates higher stress. The PSI/SF is a tool with excellent validity and reliability.
Parental Perceptions | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  A set of questionnaires developed from the previous studies will be used at T1, T2 and T3 to examine parental perceptions on the PMDs use, the training programs and children's capabilities.
Activity Log | The test will be administered on three occasions: before and after the 12-week intervention (T1 & T2) and the end of the 12-week follow up phase (T3).
  To record the training duration, locations, activities and the caregiver's feedback on the training program once every week during the intervention phase. The activity log will be mostly qualitative data that involves parents' descriptions.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Han Huang, ScD, Principal Investigator — Chang Gung University
Locations (2):
- Taiwan (2):
  - Chang Gung University, Taoyuan, Taoyuan County
  - Linkou Chang Gung Memorial Hospital, Taoyuan, Taoyuan County